CLINICAL TRIAL: NCT06740825
Title: A Phase 1, Open Label, Randomized, Parallel Drug Interaction Study to Evaluate the Effect of a CYP3A Weak Inducer Rufinamide on the Pharmacokinetics of Quizartinib in Healthy Subjects
Brief Title: Study to Assess the Effect of a CYP3A Weak Inducer Rufinamide on Quizartinib Pharmacokinetics in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC220-164
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Healthy Subjects
Keywords: Quizartinib
MeSH Terms: interventions — quizartinib; rufinamide

STUDY DESIGN:
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group A (Test) (Experimental): On Day 1 through Day 32, participants will receive an oral dose of 400-mg of rufinamide twice daily (BID). In addition, on Day 12, subjects will receive an oral single dose of 60-mg quizartinib
  Interventions: Drug: Quizartinib; Drug: Rufinamide
- Treatment Group B (Reference) (Experimental): On Day 1, participants will receive an oral dose of 60-mg quizartinib
  Interventions: Drug: Quizartinib

INTERVENTIONS:
Drug: Quizartinib — Single oral dose of 60 mg
  Other Names: VANFLYTA®
Drug: Rufinamide — Twice daily (BID) dose of 400 mg on Days 1 through 32
  Arms: Treatment Group A (Test)

SUMMARY:
This study will evaluate the effect of CYP3A weak inducer rufinamide on the pharmacokinetics (PK) of Quizartinib in healthy subjects

DETAILED DESCRIPTION:
This is a clinical pharmacology study with 2 treatment groups (Test treatment group receiving both rufinamide weak CYP3A inducer and quizartinib and Reference treatment group receiving quizartinib only) investigating the effect of rufinamide on the PK of quizartinib in healthy subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female subjects 18 to 55 years of age (inclusive), with a BMI of 18 kg/m2 to 32 kg/m2 (inclusive) at Screening.
* Has vital signs (measured after subject has been supine for at least 5 minutes) at Screening within the following ranges: heart rate: 50-100 beats per minute (bpm); systolic blood pressure (BP): 90-145 mmHg; diastolic BP: 50-95 mmHg. Out-of-range vital signs may be repeated once.
* Liver function test results (alanine aminotransferase [ALT], aspartate aminotransferase [AST], and total bilirubin [TBbil]) must be equal to or below the upper limit of normal (ULN). Hemoglobin levels must be ≥11.5 g/dL for female subjects and ≥12.5 g/dL for male subjects.
* In females, documented surgical sterilization (i.e., documented hysterectomy, bilateral tubal ligation, or bilateral salpingo-oophorectomy, Essure® with hysterosalpingogram [documentation to confirm tubal occlusion 12 weeks after procedure]), postmenopausal status for at least 1 year (follicle stimulating hormone [FSH] > 40 mIU/mL serum and estradiol <40 pg/mL [<147 pmol/L] at Screening), or agreement to have sterile male partner, or agreement to use 1 of the protocol-approved means of contraception from Screening until 7 months after the dose of quizartinib.
* In males, documented surgical sterilization, or sexual abstinence, or agreement to use 1 of the protocol-approved means of contraception from Screening until 4 months after the dose of quizartini

Key Exclusion Criteria:

* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormality) that could interfere with subject's safety, obtaining informed consent, compliance to the study procedures, or the validity of the study results.
* History of a clinically significant illness, in the opinion of the Investigator, within 4 weeks prior to administration of quizartinib.
* History or presence of an abnormal ECG, which, in the investigator's opinion, is clinically significant and/or a QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 milliseconds (ms) at Screening.
* Females who are pregnant or breastfeeding
* Laboratory results (serum chemistry, hematology, and urinalysis) outside the normal range, if considered clinically significant by the investigator. Estimated creatinine clearance (CrCl)<90 mL/min (calculated by using the Cockcroft-Gault Equation) at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter: Cmax | From day of first dose, Day 1, up to Day 33
  Cmax is defined as maximum concentration, determined directly from individual concentration-time data
Pharmacokinetic Parameter: AUClast | From day of first dose, Day 1, up to Day 33
  AUClast is defined as area under the concentration-time curve from time-zero to the time of the last quantifiable concentration; calculated using the linear up log down
Pharmacokinetic Parameter: AUCinf | From day of first dose, Day 1, up to Day 33
  AUCinf is defined as area under the concentration-time curve from time-zero extrapolated to infinity

SECONDARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) | From day of first dose, Day 1 up to the last day of Safety Follow-up, up to approximately 40 days
  TEAEs are defined as new AEs that occur after the first dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- WCT, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No